CLINICAL TRIAL: NCT00598481
Title: ADA Gene Transfer Into Hematopoietic Stem/Progenitor Cells for the Treatment of ADA-SCID
Acronym: Gene-ADA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione Telethon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STRIM-004; 15386-PRE21 (Other: IRCCS San Raffaele)
Record Dates: First submitted 2008-01-10; First posted 2008-01-22 (Estimated); Results first posted 2020-07-31 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2023-11

CONDITIONS: Immunologic Deficiency Syndromes
Keywords: SCID; gene therapy; Adenosine deaminase; retroviral vector
MeSH Terms: conditions — Immunologic Deficiency Syndromes | interventions — Genetic Therapy; Busulfan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gene Therapy (Experimental): Infusion of autologous CD34+ cells transduced with retroviral vector encoding ADA after non-myeloablative conditioning with busulfan
  Interventions: Genetic: Gene Therapy; Drug: Busulfan

INTERVENTIONS:
Genetic: Gene Therapy — Infusion of autologous CD34+ cells transduced with retroviral vector encoding ADA after non-myeloablative conditioning with busulfan
  Other Names: Gene transduced CD34+ cells; GSK2696273; Strimvelis
Drug: Busulfan — Busulfan is used for non-myeloablative conditioning

SUMMARY:
This is a phase I/II protocol to evaluate the safety and efficacy of ADA gene transfer into hematopoietic stem/progenitor cells for the treatment of adenosine deaminase (ADA)-deficiency. This condition is an autosomal recessive form of Severe Combined Immunodeficiency (SCID) characterized by impaired immune responses, recurrent infections, failure to thrive and systemic toxicity due to accumulation of purine metabolites. Transplants from an human leukocyte-antigen (HLA)-identical sibling donor is the treatment of choice, but available for a minority of patients. The use of alternative bone marrow donors or enzyme replacement therapy is associated with important drawbacks. The drug product studied in this protocol consists of autologous cluster of differentiation (CD)34+ hematopoietic stem/progenitor cells engineered ex vivo with a retroviral vector encoding the therapeutic gene ADA. The engineered CD34+ cells are infused following a nonmyeloablative conditioning with busulfan to make space in the bone marrow. The study objectives are: a) to evaluate the safety and the clinical efficacy of gene therapy, in the absence of enzyme replacement therapy; b) to evaluate the biological activity (engraftment, ADA expression) of ADA transduced CD34+ cells and their hematopoietic progeny. c) to evaluate the immunological reconstitution and purine metabolism after gene therapy.

DETAILED DESCRIPTION:
The safety of the study will be evaluated by description of all adverse events and adverse drug reactions.

The study is aimed at reaching the minimum sample size of ten patients.

ELIGIBILITY:
Inclusion Criteria:

* ADA-SCID with no HLA-identical sibling donor available
* pediatric age and at least one of the following criteria:
* inadequate immune response after PEG-ADA for > 6 months
* patients who discontinued PEG-ADA due to intolerance, allergy or auto-immunity
* patients for whom enzyme replacement therapy is not a life long therapeutic option

Exclusion Criteria:

* HIV infection
* history or current malignancy
* Patients who received a previous gene therapy treatment in the 12 months prior to receiving Strimvelis
* any other conditions dangerous for the patients according to the investigator

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2002-10-02 (Actual); Primary Completion 2011-07-10 (Actual); Study Completion 2019-06-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fondazione Telethon, Study Director — Fondazione Telethon
Locations (2):
- Investigational Site, Jerusalem, Israel
- Ospedale San Raffaele, Milan, Lombardy, Italy

REFERENCES:
- [Derived] Migliavacca M, Barzaghi F, Fossati C, Rancoita PMV, Gabaldo M, Dionisio F, Giannelli S, Salerio FA, Ferrua F, Tucci F, Calbi V, Gallo V, Recupero S, Consiglieri G, Pajno R, Sambuco M, Priolo A, Ferri C, Garella V, Monti I, Silvani P, Darin S, Casiraghi M, Corti A, Zancan S, Levi M, Cesana D, Carlucci F, Pituch-Noworolska A, AbdElaziz D, Baumann U, Finocchi A, Cancrini C, Ladogana S, Meinhardt A, Meyts I, Montin D, Notarangelo LD, Porta F, Pasquet M, Speckmann C, Stepensky P, Tommasini A, Rabusin M, Karakas Z, Galicchio M, Leonardi L, Duse M, Guner SN, Di Serio C, Ciceri F, Bernardo ME, Aiuti A, Cicalese MP. Long-term and real-world safety and efficacy of retroviral gene therapy for adenosine deaminase deficiency. Nat Med. 2024 Feb;30(2):488-497. doi: 10.1038/s41591-023-02789-4. Epub 2024 Feb 14. PMID 38355973
- [Derived] Carriglio N, Klapwijk J, Hernandez RJ, Vezzoli M, Chanut F, Lowe R, Draghici E, Nord M, Albertini P, Cristofori P, Richards J, Staton H, Appleby J, Aiuti A, Sauer AV. Good Laboratory Practice Preclinical Safety Studies for GSK2696273 (MLV Vector-Based Ex Vivo Gene Therapy for Adenosine Deaminase Deficiency Severe Combined Immunodeficiency) in NSG Mice. Hum Gene Ther Clin Dev. 2017 Mar;28(1):17-27. doi: 10.1089/humc.2016.191. PMID 28319446
- [Derived] Cicalese MP, Ferrua F, Castagnaro L, Pajno R, Barzaghi F, Giannelli S, Dionisio F, Brigida I, Bonopane M, Casiraghi M, Tabucchi A, Carlucci F, Grunebaum E, Adeli M, Bredius RG, Puck JM, Stepensky P, Tezcan I, Rolfe K, De Boever E, Reinhardt RR, Appleby J, Ciceri F, Roncarolo MG, Aiuti A. Update on the safety and efficacy of retroviral gene therapy for immunodeficiency due to adenosine deaminase deficiency. Blood. 2016 Jul 7;128(1):45-54. doi: 10.1182/blood-2016-01-688226. Epub 2016 Apr 29. PMID 27129325
- [Derived] Sauer AV, Brigida I, Carriglio N, Hernandez RJ, Scaramuzza S, Clavenna D, Sanvito F, Poliani PL, Gagliani N, Carlucci F, Tabucchi A, Roncarolo MG, Traggiai E, Villa A, Aiuti A. Alterations in the adenosine metabolism and CD39/CD73 adenosinergic machinery cause loss of Treg cell function and autoimmunity in ADA-deficient SCID. Blood. 2012 Feb 9;119(6):1428-39. doi: 10.1182/blood-2011-07-366781. Epub 2011 Dec 19. PMID 22184407
- [Derived] Cassani B, Montini E, Maruggi G, Ambrosi A, Mirolo M, Selleri S, Biral E, Frugnoli I, Hernandez-Trujillo V, Di Serio C, Roncarolo MG, Naldini L, Mavilio F, Aiuti A. Integration of retroviral vectors induces minor changes in the transcriptional activity of T cells from ADA-SCID patients treated with gene therapy. Blood. 2009 Oct 22;114(17):3546-56. doi: 10.1182/blood-2009-02-202085. Epub 2009 Aug 3. PMID 19652199
- [Derived] Sauer AV, Mrak E, Hernandez RJ, Zacchi E, Cavani F, Casiraghi M, Grunebaum E, Roifman CM, Cervi MC, Ambrosi A, Carlucci F, Roncarolo MG, Villa A, Rubinacci A, Aiuti A. ADA-deficient SCID is associated with a specific microenvironment and bone phenotype characterized by RANKL/OPG imbalance and osteoblast insufficiency. Blood. 2009 Oct 8;114(15):3216-26. doi: 10.1182/blood-2009-03-209221. Epub 2009 Jul 24. PMID 19633200
- [Derived] Aiuti A, Cattaneo F, Galimberti S, Benninghoff U, Cassani B, Callegaro L, Scaramuzza S, Andolfi G, Mirolo M, Brigida I, Tabucchi A, Carlucci F, Eibl M, Aker M, Slavin S, Al-Mousa H, Al Ghonaium A, Ferster A, Duppenthaler A, Notarangelo L, Wintergerst U, Buckley RH, Bregni M, Marktel S, Valsecchi MG, Rossi P, Ciceri F, Miniero R, Bordignon C, Roncarolo MG. Gene therapy for immunodeficiency due to adenosine deaminase deficiency. N Engl J Med. 2009 Jan 29;360(5):447-58. doi: 10.1056/NEJMoa0805817. PMID 19179314
- [Derived] Cassani B, Mirolo M, Cattaneo F, Benninghoff U, Hershfield M, Carlucci F, Tabucchi A, Bordignon C, Roncarolo MG, Aiuti A. Altered intracellular and extracellular signaling leads to impaired T-cell functions in ADA-SCID patients. Blood. 2008 Apr 15;111(8):4209-19. doi: 10.1182/blood-2007-05-092429. Epub 2008 Jan 24. PMID 18218852

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The Pivotal study enrolled 12 participants.
Groups:
- Gene Therapy: Infusion of autologous cluster of differentiation (CD)34+ cells transduced with retroviral vector encoding ADA after non-myeloablative conditioning with busulfan
Period: Baseline
Arm/Group | Gene Therapy
Started | 12
Completed | 12
Not Completed | 0
Period: Treatment
Arm/Group | Gene Therapy
Started | 12
Completed | 11
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Population: The Intention to Treat (ITT) Population included all subjects who were treated with gene therapy and had at least 1 post-therapy evaluation during the 0-3year follow-up.
Groups:
- Gene Therapy (Pivotal): Infusion of autologous cluster of differentiation (CD)34+ cells transduced with retroviral vector encoding ADA after non-myeloablative conditioning with busulfan
Arm/Group | Gene Therapy (Pivotal)
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 12
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 2.38 [0.5 to 6.1]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Italy | 12

OUTCOME MEASURES:

1. Primary Outcome: Survival
Description: From post-treatment to up to 3 years
Time Frame: baseline to 3 years post gene therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Gene Therapy (Pivotal)
Number analyzed (Participants) | 12
Participants | 12

2. Secondary Outcome: Rate of Severe Infections
Description: Severe infections were defined as those that required hospitalization or those that prolonged hospitalization. The rate of infection was estimated as number of severe infections over person-years of observation (free from severe infections) before and after treatment administration. The first 3 months after gene therapy were not considered in the post-gene therapy analysis, because all subjects were hospitalized during this period.
Time Frame: Before Treatment and 3-months post-treatment up to 3 years
Measure: Number; unit: Severe Infections per person year
Groups:
- Severe Infections (Before Gene Therapy): This is the rate of severe infections prior to gene therapy.
- Severe Infections (After Gene Therapy): This is the rate of severe infections post gene therapy, taken from 3 months post gene therapy to three years post gene therapy.
Arm/Group | Severe Infections (Before Gene Therapy) | Severe Infections (After Gene Therapy)
Number analyzed (Participants) | 12 | 12
Severe Infections per person year | 1.1 | 0.429
Statistical Analysis 1: Comparison: Severe Infections (Before Gene Therapy) vs Severe Infections (After Gene Therapy); Test type: Superiority; p = 0.005, One-sided Poisson-regression

3. Secondary Outcome: CD3+ Cell Counts
Description: T-lymphocyte counts (CD3+): mean T-lymphocyte at Baseline and 3 years post gene therapy. Samples were taken from peripheral venous whole blood and tested by cytofluorometry; values are means (10^6/L).
Time Frame: baseline up to 3 years post gene therapy
Population: Only subjects with available data at each visit were included in the analysis
Measure: Geometric Mean (95% Confidence Interval); unit: 10^6 cells/L
Groups:
- Gene Therapy ITT Population: Included all subjects who were treated with gene therapy and had at least 1 year post therapy during the 0-3 year follow up
Arm/Group | Gene Therapy ITT Population
Number analyzed (Participants) | 12
10^6 cells/L
  Baseline: number analyzed (Participants) | 11
  Baseline | 112.5 [39.4 to 321]
  Year 1 | 348.3 [194.5 to 623.8]
  Year 2: number analyzed (Participants) | 11
  Year 2 | 633 [482.9 to 829.8]
  Year 3: number analyzed (Participants) | 11
  Year 3 | 831.1 [596.7 to 1157.6]
Statistical Analysis 1: Comparison: Gene Therapy ITT Population; Test type: Superiority; p = 0.003, Mixed Model Repeated Measures — P value related to geometric mean ratio at 1 year post gene therapy compared to baseline; Geometric mean ratio = 3.0, 95% CI 2-sided [1.45 to 6.19]
Statistical Analysis 2: Comparison: Gene Therapy ITT Population; Test type: Superiority; p < 0.001, Mixed Model Repeated Measures — P value related to geometric mean ratio at 2 years post gene therapy compared to baseline; Geometric mean ratio = 5.4, 95% CI 2-sided [2.63 to 11.25]
Statistical Analysis 3: Comparison: Gene Therapy ITT Population; Test type: Superiority; p < 0.001, Mixed Model Repeated Measures — P value related to geometric mean ratio at 3 years post gene therapy compared to baseline; Geometric mean ratio = 6.5, 95% CI 2-sided [3.08 to 13.64]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from pre-treatment through year 3, post gene therapy
Arm/Group | Gene Therapy (Pivotal)
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 10/12
Other Adverse Events (participants affected / at risk) | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gene Therapy (Pivotal) (N=12)
Device related infection (Infections and infestations) | 5
Gastroenteritis (Infections and infestations) | 2
Esptein-Barr virus infection (Infections and infestations) | 1
Respiratory Tract Infection (Infections and infestations) | 1
Upper Respiratory tract infection (bacterial) (Infections and infestations) | 1
Urinary Tract Infection (Infections and infestations) | 1
Varicella (Infections and infestations) | 1
Neutropenia (Blood and lymphatic system disorders) | 2
Aplastic anemia (Blood and lymphatic system disorders) | 1
Autoimmune thrombocytopenia (Blood and lymphatic system disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 1
Autoimmune hepatitis (Hepatobiliary disorders) | 1
Lipofibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hypertension (Vascular disorders) | 1
Guillian-Barre Syndrome (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Gene Therapy (Pivotal) (N=12)
Autoimmune haemolytic anemia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 4
Eosinophilia (Blood and lymphatic system disorders) | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Rhinitis (Infections and infestations) | 8
Device related infection (Infections and infestations) | 2
Upper respiratory tract infection (Infections and infestations) | 5
Gastroenteritis (Infections and infestations) | 2
Oral candidiasis (Infections and infestations) | 4
Bronchitis (Infections and infestations) | 3
Escherichia urinary tract infection (Infections and infestations) | 3
Nasopharyngitis (Infections and infestations) | 2
Upper respiratory tract infection bacterial (Infections and infestations) | 3
Urinary traction infection pseudomonal (Infections and infestations) | 3
Varicella (Infections and infestations) | 2
Hemophilus infection (Infections and infestations) | 2
Otitis media (Infections and infestations) | 2
Respiratory tract infection (Infections and infestations) | 1
Gastroenteritis norovirus (Infections and infestations) | 1
Gingivitis (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Otitis media acute (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Pneumococcal infection (Infections and infestations) | 1
Respiratory syncytial virus infection (Infections and infestations) | 1
Skin infection (Infections and infestations) | 1
Staphylococcal infection (Infections and infestations) | 1
Streptococcal infection (Infections and infestations) | 1
Tinea capitis (Infections and infestations) | 1
Urinary tract infection enterococcal (Infections and infestations) | 1
Viral diarrhea (Infections and infestations) | 1
Computerized tomogram thorax abnormal (Investigations) | 3
Hepatic enzyme increased (Investigations) | 5
Blood immunoglobulin E increased (Investigations) | 2
Electrophoresis protein abnormal (Investigations) | 2
Blood alkaline phosphatase increased (Investigations) | 2
Pseudomonas test positive (Investigations) | 1
Tympanometry abnormal (Investigations) | 2
Weight decreased (Investigations) | 2
Adenovirus test positive (Investigations) | 1
Bacterial test positive (Investigations) | 1
Clostridium test positive (Investigations) | 1
Pulmonary function test abnormal (Investigations) | 1
Serum ferritin decreased (Investigations) | 1
Spirometry abnormal (Investigations) | 1
Staphylococcus test positive (Investigations) | 1
Total lung capacity decreased (Investigations) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Bronchial wall thickening (Respiratory, thoracic and mediastinal disorders) | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Nasal turbinate hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary calcification (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 3
Dermatitis (Skin and subcutaneous tissue disorders) | 2
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 2
Skin ulcer (Skin and subcutaneous tissue disorders) | 1
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 1
Eczema nummular (Skin and subcutaneous tissue disorders) | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1
Lichen planus (Skin and subcutaneous tissue disorders) | 1
Petechiae (Skin and subcutaneous tissue disorders) | 1
Scab (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 2
Phimosis (Congenital, familial and genetic disorders) | 2
Cryptorchism (Congenital, familial and genetic disorders) | 1
Congenital genital malformation (Congenital, familial and genetic disorders) | 1
Micropenis (Congenital, familial and genetic disorders) | 1
Reproductive tract hypoplasia, male (Congenital, familial and genetic disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Enteritis (Gastrointestinal disorders) | 2
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1
Dental caries (Gastrointestinal disorders) | 1
Oral disorder (Gastrointestinal disorders) | 1
Developmental delay (General disorders) | 1
Adverse drug reaction (General disorders) | 1
Device occlusion (General disorders) | 1
Cerebral hematoma (Nervous system disorders) | 1
Psychomotor hyperactivity (Nervous system disorders) | 1
Speech disorder (Nervous system disorders) | 1
Hepatomegaly (Hepatobiliary disorders) | 1
Autoimmune hepatitis (Hepatobiliary disorders) | 1
Gallbladder cholesterolosis (Hepatobiliary disorders) | 1
Hepatic fibrosis (Hepatobiliary disorders) | 1
Hepatic lesion (Hepatobiliary disorders) | 1
Bone development abnormal (Musculoskeletal and connective tissue disorders) | 2
Hypothyroidism (Endocrine disorders) | 2
Tibia fracture (Injury, poisoning and procedural complications) | 1
Wound (Injury, poisoning and procedural complications) | 1
Food aversion (Psychiatric disorders) | 1
Deafness bilateral (Ear and labyrinth disorders) | 2
Deafness (Ear and labyrinth disorders) | 1
Middle ear inflammation (Ear and labyrinth disorders) | 1
Amblyopia (Eye disorders) | 1
Hypermetropia (Eye disorders) | 1
Myopia (Eye disorders) | 1
Refraction disorder (Eye disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Pulmonary valve stenosis (Cardiac disorders) | 1
Sinus arrhythmia (Cardiac disorders) | 1
Wandering pacemaker (Cardiac disorders) | 1
Acquired phimosis (Reproductive system and breast disorders) | 2
Perineal erythema (Reproductive system and breast disorders) | 1
Hemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lipofibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pyogenic granuloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Anaphylactic reaction (Immune system disorders) | 1
Hypertonic bladder (Renal and urinary disorders) | 1
Acidosis (Metabolism and nutrition disorders) | 1
Aspergillis infection (Infections and infestations) | 1
Campylobacter infection (Infections and infestations) | 1
Candida infection (Infections and infestations) | 2
Catheter site infection (Infections and infestations) | 1
Clostridium difficile colitis (Infections and infestations) | 1
Clostridium difficile infection (Infections and infestations) | 1
Ear infection (Infections and infestations) | 2
Escherichia sepsis (Infections and infestations) | 1
Fungal skin infection (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Staphylococcal sepsis (Infections and infestations) | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 4
Autoimmune thrombocytopenia (Blood and lymphatic system disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 4
Pyrexia (General disorders) | 4
Epstein-Barr virus infection (Infections and infestations) | 1
Respiratory Tract Infection, bacterial (Infections and infestations) | 1
Urinary Tract Infection (bacterial) (Infections and infestations) | 2
Hypertension (Vascular disorders) | 3
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less